CLINICAL TRIAL: NCT02528110
Title: A Phase II Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in the Treatment of Locally Advanced Gastric Cancer During Radical Gastrectomy
Brief Title: Radical Gastrectomy and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Locally Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Cancer Center of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU_HIPEC
Record Dates: First submitted 2015-08-16; First posted 2015-08-19 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Malignant Neoplasm of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radical gastrectomy without HIPEC (Sham Comparator): Patients will be treated with a D2 radical gastrectomy for locally advanced gastric cancer and postoperative chemotherapy (SOX or XELOX)
  Interventions: Procedure: D2 radical gastrectomy; Other: SOX postoperative chemotherapy; Other: XELOX postoperative chemotherapy
- Radical gastrectomy with HIPEC (Experimental): Patients will be treated with a D2 radical gastrectomy for locally advanced gastric cancer and HIPEC with paclitaxel and 5-Fu and postoperative chemotherapy (SOX or XELOX)
  Interventions: Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC); Procedure: D2 radical gastrectomy; Other: SOX postoperative chemotherapy; Other: XELOX postoperative chemotherapy

INTERVENTIONS:
Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) — Normal saline 3000ml-4000ml, Paclitaxel 75mg/m2, 5-Fu 15mg/m2, 43°C, 60min.
  Arms: Radical gastrectomy with HIPEC
Procedure: D2 radical gastrectomy — radical gastrectomy with D2 lymphadenectomy
Other: SOX postoperative chemotherapy — Oxaliplatin 130mg/m2 d1, Tegafur,Gimeracil and Oteracil Porassium Capsules 60mg, d1-14.
Other: XELOX postoperative chemotherapy — Oxaliplatin 130mg/m2 d1, Capecitabine 1000mg/m2 d1-14.

SUMMARY:
The efficacy of HIPEC in prevention of local recurrence, distant metastasis or peritoneal metastasis in locally advanced gastric cancer is not definite. The hypothesis of the trial is that radical gastrectomy plus HIPEC is superior to only radical gastrectomy in terms of overall survival.

DETAILED DESCRIPTION:
To determine the efficacy of HIPEC in the treatment of locally advanced gastric cancer, patients are randomized into HIPEC group and control group. In HIPEC group, the patients undergo radical gastrectomy with D2 lymphadenectomy and HIPEC with paclitaxel and 5-Fu. Patients in the control group just undergo radical gastrectomy with D2 lymphadenectomy. Patients in both groups receive 6 cycles of postoperative chemotherapy (SOX or XELOX) and are followed up for 5 years or until death.

The trial is designed as a prospective, randomized, open, multicenter and parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of locally advanced gastric cancer.
* No evidence of distant metastases or peritoneal metastases.
* Preoperative examination (CT/MRI) demonstrated resectable gastric cancer with T3-T4 stage.
* Eligible for radical gastrectomy with D2 lymphadenectomy.
* Have not received cytotoxic chemotherapy or radiotherapy.
* Written informed consent is obtained prior to commencement of trial treatment.

Exclusion Criteria:

* Existence of distant metastasis or peritoneal metastasis during surgery (M1).
* Any previous chemotherapy or radiotherapy
* Active systemic infections
* Inadequate cardiac function, renal function, liver function or bone marrow function at the beginning of the trial.
* Female patients who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  From the date of surgery to the date of death or to the end of follow-up

SECONDARY OUTCOMES:
progression-free survival | 5 years
distant metastasis rate | 5 years
peritoneal metastasis rate | 5 years
local recurrence rate | 5 years
complication rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China